CLINICAL TRIAL: NCT03747926
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 705564 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: This Study is Done in Healthy Japanese Volunteers. It Looks at How Different Doses of BI 705564 Are Taken up in the Body and How Well They Are Tolerated
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Substance discontinued.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1408-0005
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 705564 (Experimental)
  Interventions: Drug: BI 705564
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 705564 — single-rising oral dose
  Arms: BI 705564
Drug: Placebo — single-rising oral dose
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 705564 in healthy male subjects following oral administration of single rising doses.

A secondary objective is the exploration of the PK including dose proportionality of BI 705564 after single dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR), Respiratory Rate (RR), body temperature), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 20 to 50 years (incl.) at screening
* Body Mass Index (BMI) of 18.5 to 25.0 kg/m2 (incl.) at screening
* Signed and dated written informed consent in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male subject who agree to minimize the risk of female partners becoming pregnant by fulfilling any of the following criteria starting from at least 30 days before the first administration of trial medication and until 90 days after the trial completion:

  * Use of adequate contraception, e.g., any of the following methods plus condom:

    --- combined oral contraceptives, intrauterine device.
  * Vasectomised (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilised (including hysterectomy) of the subject's female partner

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic BP outside the range of 90 to 140 mmHg, diastolic BP outside the range of 50 to 90 mmHg, or pulse rate (PR) outside the range of 45 to 90 beats per minute (bpm) at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance at screening
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders, including but not limited to mood disorders and any history of suicidality
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including human immunodeficiency virus (HIV), viral hepatitis, syphilis and/or tuberculosis or evidence of tuberculosis infection as defined by positive QuantiFERON TB-Gold (or T-SPOT) test. (Subject with positive Hepatitis B core antibody will not allowed to participate in this study)
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days or 5 half-lives, whichever is longer prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 200 mL within 30 days or 400 mL within 12 weeks prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 msecond) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Subjects who, in the investigator's judgement, are perceived as having an increased risk of bleeding, e.g., history of haemorrhagic disorders, clinical relevant petechial bleeding, occult blood in faeces, haematuria in repeated urine tests, trauma or surgery within the last month, planned surgery during trial participation, history of arteriovenous malformation or aneurysm, history of gastroduodenal ulcer disease or gastrointestinal haemorrhage, history of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intraarticular bleeding, use of drugs that may interfere with haemostasis during trial conduct (e.g., acetylic salicylic acid or other non-steroidal anti-inflammatory drugs)
* Repeated absolute B cell (CD19+) counts below 40/μL at screening
* Repeated platelet counts below 100 cells/nL (10.0×104/μL) at screening
* Serum potassium below normal range at screening
* A history or current clinical signs of acute pancreatitis

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-05 (Estimated); Primary Completion 2019-08-12 (Estimated); Study Completion 2019-09-02 (Estimated)

PRIMARY OUTCOMES:
Number [N (%)] of subjects with drug-related Adverse Events (AEs) | Up to day 7

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 72 hours
Cmax (maximum measured concentration of the analyte in plasma) | Up to 72 hours

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing